CLINICAL TRIAL: NCT04673162
Title: A Randomized, Multicentre, Double-blind Study to Evaluate the Efficacy of High-dose Administration of Methylprednisolone in Addition to Standard Treatment, in SARS-CoV2 (COVID-19) Pneumonia Patients
Brief Title: Evaluation of the Efficacy of High Doses of Methylprednisolone in SARS-CoV2 ( COVID-19) Pneumonia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-MP-COVID-19
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Covid19; Methylprednisolone
MeSH Terms: conditions — COVID-19 | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Randomized, multicentric, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A SOC plus MP (Experimental): Standard treatment (currently desamethasone 6mg/daily for 10 days) plus Methylprednisolone 1gr daily iv on days 1,2,3
  Interventions: Drug: Methylprednisolone, Placebo
- B SOC plus Pb (Active Comparator): Standard treatment (currently desamethasone 6mg/daily for 10 days) plus Placebo
  Interventions: Drug: Methylprednisolone, Placebo

INTERVENTIONS:
Drug: Methylprednisolone, Placebo — iv administration
  Other Names: Standard treatment

SUMMARY:
This double blind, randomized study is aiming to evaluate the efficacy of three doses (1gr/day) of methylpredisolone added to standard therapy in patients, with documented COVID-19 pneumonia, requiring hospitalization but not mechanical ventilation.

DETAILED DESCRIPTION:
Patients recently hospitalized for the treatment of documented COVID-19 pneumonia who do not require invasive ventilation will be randomized (1:1) to receive current standard treatment, which may include desamethasone and oxygen, with methylprenisolone 1gr daily iv for 3 consecutive days or standard treatment alone.

Efficacy measures will be time to recovery (discharge from hospital), invasive ventilation prevention and survival.

Patients safety will be evaluated throughout the all study period.

ELIGIBILITY:
Inclusion Criteria:

1. age = 18 years;
2. Informed consent for participation in the study and for data processing;
3. Molecular diagnosis with Polymerase Chain Reaction (PCR) test of Sars-CoV2 infection;
4. Hospitalization in a specialist ward for Covid-19 patient care (eg., Infectious Diseases, Pulmonology or Internal Medicine);
5. Need for supplemental oxygen in any delivery mode with the exception of invasive mechanical ventilation;
6. PaO2 / FiO2 between 100 and 300 mmHg.
7. Clinical / instrumental diagnosis (high resolution chest CT scan or chest x-ray or lung ultrasound) of interstitial pneumonia for no more than three days;
8. Serum CRP greater than 5 mg / dL;
9. Interval from onset of SARS-CoV2 infection symptoms to randomization> 5 days-

Exclusion Criteria:

1. Invasive mechanical ventilation;
2. Presence of shock or concomitant organ failure that requires admission to the Intensive Care Unit;
3. Pregnancy or breastfeeding;
4. Severe heart or kidney failure;
5. Known hypersensitivity to methylprednisolone, to dexamethasone or to an exception;
6. Diabetes not compensated according to the doctor's judgment;
7. Other clinical conditions that contraindicate Methylprednisolone and cannot be treated or resolved according to the doctor's judgment;
8. Steroid bolus therapy in the week prior to enrollment for the study;
9. Enrollment in another clinical trial;
10. Patient already randomized in this study-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | 30 days since randomisation
  the interval between randomization and discharge from the hospital without the need for supplemental oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Costantini, MD, Study Chair — AUSL-IRCCS di Reggio Emilia
Locations (20):
- Italy (20):
  - UO di Malattie Infettive, Azienda Sociosanitaria Ligure 1, Sanremo, Imperia
  - SOC di Pneumologia, Az. Osp. S. Antonio e Biagio e C. Arrigo, Alessandria
  - UO di Pneumologia, Ospedale San Donato, Arezzo
  - UO di Malattie Infettive, Policlinico Sant'Orsola Malpighi, Bologna
  - UO di Pneumologia e Terapia Intensiva Respiratoria, Policlinico Sant' Orsola Malpighi, Bologna
  - Reparto di Malattie Infettive, Comprensorio Sanitario di Bolzano- Az. Sanitaria Alto Adige, Bolzano
  - SOC di Malattie Infettive, ASST di Cremona, Cremona
  - SOC di Malattie Infettive, AOU Careggi, Florence
  - UOC di Pneumologia, IRCCS Ospedale Policlinico San Martino, Genova
  - SC di Malattie Infettive,Ospedale Sant'Andrea - Az. Sociosanitaria Ligure 5, La Spezia
  - UO Malattie Infettive, Azienda Ospedaliera Universitaria- Policlinico di Modena, Modena
  - UO Clinica Pneumologica - Ospedale "San Gerardo" - ASST di Monza, Monza
  - UO Terapia Anestesia e Rianimazione - Ospedale "San Gerardo" - ASST di Monza, Monza
  - UO di Malattie Infettive, Ospedale Guglielmo da Saliceto - AUSL di Piacenza, Piacenza
  - UO di Pneumologia, Ospedale Guglielmo da Saliceto - AUSL di Piacenza, Piacenza
  - SOC di Malattie Infettive - AUSL-IRCCS di Reggio Emilia, Reggio Emilia
  - SOC di Pneumologia - AUSL-IRCCS di Reggio Emilia, Reggio Emilia
  - SOC di Reumatologia, AUSL- IRCCS di Reggio Emilia, Reggio Emilia
  - UOC di Malattie Infettive - Azienda Unità Locale Socio Sanitaria n. 2, Treviso
  - UO di Pneumologia, Azienda Ospedaliera Universitaria Integrata, Verona

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as the main results have been published
Access Criteria: publication reviewers

REFERENCES:
- [Derived] Salvarani C, Massari M, Costantini M, Merlo DF, Mariani GL, Viale P, Nava S, Guaraldi G, Dolci G, Boni L, Savoldi L, Bruzzi P, Turra C, Catanoso M, Marata AM, Barbieri C, Valcavi A, Franzoni F, Cavuto S, Mazzi G, Corsini R, Trapani F, Bartoloni A, Barisione E, Barbieri C, Burastero GJ, Pan A, Inojosa W, Scala R, Burattini C, Luppi F, Codeluppi M, Tarek KE, Cenderello G, Salio M, Foti G, Dongilli R, Bajocchi G, Negri EA, Ciusa G, Fornaro G, Bassi I, Zammarchi L, Aloe T, Facciolongo N. Intravenous methylprednisolone pulses in hospitalised patients with severe COVID-19 pneumonia: a double-blind, randomised, placebo-controlled trial. Eur Respir J. 2022 Oct 20;60(4):2200025. doi: 10.1183/13993003.00025-2022. Print 2022 Oct. PMID 35361632